CLINICAL TRIAL: NCT05114928
Title: Correlation Between Changes in Corneal Asphericity and Progression of Keratoconus in Children
Brief Title: Correlation Between Q-value Changes and Progression of Pediatric Keratoconus.
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Lecturer of Ophthalmology, Benha University
Other Study IDs: RC-10-7-01
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Keratoconus; Collagen Diseases; Corneal Disease
Keywords: corneal asphericity; corneal collagen cross-linking; Q-value; Pediatric keratoconus; Trans-epithelial
MeSH Terms: conditions — Keratoconus; Collagen Diseases; Corneal Diseases | interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Progression Group (P-group): Eyes that showed progression of the disease after trans-epithelial corneal collagen cross-linking during the 5 years of follow-up, (number of eyes = 7 eyes).
  Interventions: Procedure: Transepithelial Corneal Collagen Cross-linking; Diagnostic Test: Scheimpflug camera
- No Progression Group (NP-group): Eyes that showed no progression of the disease after trans-epithelial corneal collagen cross-linking during the 5 years of follow-up, (number of eyes = 11 eyes).
  Interventions: Procedure: Transepithelial Corneal Collagen Cross-linking; Diagnostic Test: Scheimpflug camera

INTERVENTIONS:
Procedure: Transepithelial Corneal Collagen Cross-linking — Bilateral Transepithelial Corneal Collagen Cross-linking was done for all subjects using power of 9mW/cm2 at 55mm from the cornea for 10 minutes, with a total energy of 5.4j/cm2 using the (CCL VARIO, PESCHKE Trade GmbH, Huenenberg Switzerland), in the period between January 2016 to August 2016.
  Other Names: TE-CXL
Diagnostic Test: Scheimpflug camera — Pentacam (OCULUS Optikgeräte GmbH, Wetzlar, Germany) was done for all subjects at baseline and annually after TE-CXL till 5 years of follow-up.
  Other Names: Pentacam

SUMMARY:
Keratoconus is a progressive corneal disease characterized by asymmetric corneal thinning and structural changes in corneal collagen which leads to decrease in visual acuity due to myopic shift, irregular astigmatism or corneal scarring. Early detection of the disease in children aids in halting the progression and improve their quality of life. There is no consensus regarding the progression criteria of the disease, we aimed to assess the changes in corneal asphericity in children after corneal collagen crosslinking and investigate any possible correlation with progression criteria widely used.

DETAILED DESCRIPTION:
The Keratoconus progression is defined as increasing by 1.0 diopter (D) or more in the maximum keratometry (Kmax), progressive deterioration in Minimal Corneal Thickness is also associated with KC progression, other methods have been investigated to confirm KC progression such as changes in manifest refraction, unaided visual acuity (UAVA), BCVA, posterior keratometric data and higher order aberrations (HOA) which are altered in KC and can aid to confirm disease progression. Q-value (a coefficient of corneal asphericity) reflects the shape of the cornea, its refractive power, and spherical aberration. The mean Q-value in normal cornea is -0.26 ± 0.18, the severity of KC and the Q-value are inversely related.

Mean Q-value in KC at 8mm zone is -0.84 and -1.10 for anterior and posterior corneal surfaces, respectively. Until now, no precise criteria of KC progression especially in cases had undergone previous trans-epithelial corneal collagen cross-linking (TE-CXL) to halt the progression of the disease. In the present study we aimed to analyze the correlation between the changes in Q-value and progression of the KC in children had undergone bilateral TE-CXL.

ELIGIBILITY:
Inclusion Criteria:

Children that were diagnosed as bilateral progressive KC (stage I-III, according to amsler classification, Kmax change >1D between 2 scanning with at least 2 months apart), and their age were less than 16 years old at time of TE-CXL, topographic parameters were Kmax 47-60D and MCT more than 400μm.

Exclusion Criteria:

Eyes with central corneal scarring, amblyopic eyes, and other corneal pathologies that may alter Pentacam scanning.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This retrospective observational study was performed at Ophthalmology department, Benha University, EGYPT using the medical records of 9 children diagnosed as bilateral progressive KC that was confirmed by Pentacam according to amsler criteria, patients had undergone bilateral TE-CXL in the period from January 2016 to August 2016 and completed annual visits till 5 years of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-10-09 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Changes in corneal asphericity (Q-value) in all subjects. | Baseline and annually after TE-CXL till 5 years of follow-up
  Evaluate the changes in Q-value after Trans-epithelial corneal collagen cross-linking (TE-CXL) using pentacam.

SECONDARY OUTCOMES:
Correlation between Q-value changes and disease progression in both groups. | Baseline and annually after TE-CXL till 5 years of follow-up
  Correlation between the changes in Q-value in different corneal zones and maximum keratometry and minimal corneal thickness in both groups over 5 years of follow-up.
The Q-value as a predictive value in keratoconus progression. | Baseline and annually after TE-CXL till 5 years of follow-up
  The possibility of using the Q-value parameters as a predictive values to confirm keratoconus progression in children.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Tabl, MD, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy Tabl, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Undecided